CLINICAL TRIAL: NCT07002879
Title: Comparison Of Ultrasound-guided Dry Needling and Platelet-rich Plasma Administration in the Treatment of Refractory Lateral Epicondylitis
Brief Title: Ultrasound-Guided Dry Needling vs PRP for Refractory Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Yusuf Kıratlıoğlu, Ankara University, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: İ07-436-22
Record Dates: First submitted 2025-05-25; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2022-01

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dry needle (Active Comparator): An 18-gauge needle was first used to fenestrate the common extensor tendon and lateral periosteum. Once adequate anesthesia was confirmed, an 18-gauge needle was inserted along the tendon's longitudinal axis (without exiting the skin) and advanced in a "peppering" motion 40 to 50 passes from superficial to deep layers over approximately two minutes.
  Interventions: Procedure: dry needle
- platelet rich plasma injection (Active Comparator): A 15 mL peripheral blood sample was drawn and centrifuged at 3 000 rpm for 3 minutes. Approximately 2 mL of PRP was aspirated directly from the buffy coat and injected into the epicondylar region under ultrasound guidance.
  Interventions: Procedure: Platelet Rich Plasma

INTERVENTIONS:
Procedure: dry needle — An 18-gauge needle was first used to fenestrate the common extensor tendon and lateral periosteum. Once adequate anesthesia was confirmed, an 18-gauge needle was inserted along the tendon's longitudinal axis (without exiting the skin) and advanced in a "peppering" motion 40 to 50 passes from superficial to deep layers over approximately two minutes
  Arms: dry needle
Procedure: Platelet Rich Plasma — A 15 mL peripheral blood sample was drawn and centrifuged at 3 000 rpm for 3 minutes. Approximately 2 mL of PRP was aspirated directly from the buffy coat and injected into the epicondylar region under ultrasound guidance.
  Arms: platelet rich plasma injection

SUMMARY:
This single-center, randomized, prospective study was conducted between January 2022 and September 2023 with ethics committee approval. Adults aged 18-65 with a clinical diagnosis of lateral epicondylitis-characterized by lateral elbow pain exacerbated by resisted wrist or middle finger extension-and who had not responded to at least six weeks of conservative treatment were included. Exclusion criteria included cervical disc disease, nerve entrapment, arthrosis, uncontrolled metabolic disorders, bleeding disorders, prior elbow surgery or injection, pregnancy, cognitive impairment, or compromised skin at the injection site. A G*Power sample size calculation determined that at least 50 patients were needed.

Participants were randomly assigned to two groups: 25 received ultrasound-guided dry needling and 25 received platelet-rich plasma (PRP) injections. All participants gave informed consent, and the study adhered to the Declaration of Helsinki. Baseline demographic and clinical data were collected, and the diagnosis was confirmed using Mills, Maudsley, and Thomsen tests, along with grip-strength assessment. Pain and function were evaluated using the PRTEE, Visual Analog Scale (VAS), and QuickDASH questionnaires at baseline, and at 1, 3, and 6 months post-treatment.

Ultrasound imaging was used to identify tendinopathic changes. Local anesthesia was administered with 2 mL of prilocaine.

In the dry needling group, an 18-gauge needle was used to fenestrate the tendon with 40-50 passes in a "peppering" motion under continuous ultrasound guidance.

In the PRP group, 15 mL of blood was drawn, centrifuged, and approximately 2 mL of PRP was injected into the lesion under ultrasound guidance.

After the procedure, patients were advised to apply ice, perform passive stretching, avoid lifting heavy objects, and refrain from NSAID use for two weeks. Gradual return to normal activities was encouraged thereafter to restore full elbow function.

ELIGIBILITY:
Inclusion Criteria: 18 and 65 years of age, having a clinical diagnosis of lateral epicondylitis based on localized lateral elbow pain exacerbated by resisted wrist or middle finger extension and tenderness over the lateral epicondyle on physical examination, and failure to respond to at least six weeks of conservative treatment.

-

Exclusion Criteria:the presence of cervical discopathy or upper extremity nerve entrapment, radiocapitellar arthrosis, uncontrolled metabolic diseases (hypothyroidism, diabetes), bleeding diathesis, a history of previous elbow injection or surgery, pregnancy or lactation, cognitive impairment, and skin compromise at the injection site

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 1-3-6 months
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire | 1-3-6 months
Patient-Rated Tennis Elbow Evaluation | 1-3-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No